CLINICAL TRIAL: NCT01521364
Title: The Pharmacokinetic Effect of Clarithromycin on the AUC0-12h of Linezolid in Multidrug-resistant and Extensively Drug-resistant Tuberculosis (MDR/XDR-TB) Patients
Brief Title: Drug Interaction Study Between Linezolid and Clarithromycin in Tuberculosis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, JWC Alffenaar, PhD, Pharm D, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL35534.042.11; 2011-000513-39 (EudraCT Number)
Record Dates: First submitted 2011-09-13; First posted 2012-01-30 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-05

CONDITIONS: Multidrug-resistant Tuberculosis; Extensively Drug-resistant Tuberculosis
Keywords: pharmacokinetic; drug-interaction; linezolid; clarithromycin; Mycobacterium tuberculosis
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis | interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0mg, 250mg, and 500mg claritromycin (Other): Patients receive 300mg linezolid twice a day during entire study. After one week, 250mg claritromycin once daily is added for a duration of two weeks.
  After another two weeks, 250mg claritromycin is replaced by 500mg claritromycin once daily for another two weeks.
  After this, there is a wash-out period of one week during which no claritromycine is administered.
  Interventions: Drug: Addition of different doses of clarithromycin.

INTERVENTIONS:
Drug: Addition of different doses of clarithromycin. — At week 1, 250mg clarithromycin once a day will be added to linezolid therapy during two weeks.
  At week 3, 500mg clarithromycin once a day will be added to linezolid therapy during to weeks.
  Other Names: Clarithromycin, 250/500mg (Pharmachemie) RVG 029081/029082

SUMMARY:
Future patients might benefit from a combination of linezolid (LIN) and clarithromycin (CLA) in the treatment of Multidrug-resistant and Extensively Drug-resistant Tuberculosis (MDR/XDR-TB) due to possible synergistic activity as shown in in vitro experiments in different Mycobacteria strains. The investigators observed increased LIN serum levels in three cases after combining LIN and CLA of which the investigators described one in a case report (Bolhuis et al). The investigators suggest to conduct a prospective pharmacokinetic study in MDR- and XDR-TB patients to quantify the above described interaction between LIN and CLA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Signed informed consent
* Diagnosis of MDR/XDR-TB confirmed with standard microbiological criteria (culture-based, molecular or both)
* Treatment with linezolid 300mg twice daily per os.

Exclusion Criteria:

* Hypersensitivity to: linezolid, clarithromycin, erythromycin, or any macrolide antibiotics, or any of the excipients of linezolid or clarithromycin.
* Concomitant use with astemizole, cisapride, ergotamine derivatives (dihydroergotamine, ergotamine), monoamine oxidase inhibitors (phenelzine, isocarboxazid, selegiline, or moclobemide), pimozide, or terfenadine.
* Pregnancy or breast-feeding.
* Hypokalemia
* Concomitant use of other P-gp inhibitors/inducers, e.g. amiodarone, verapamil, digoxin, tipranavir/ritonavir, lovastatin, tariquidar, itraconazole, dipyridamol, erythromycin, ritonavir, quinidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem C Alffenaar, PhD, PharmD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Tuberculosis Center Beatrixoord, Haren, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Bolhuis MS, van Altena R, van Soolingen D, de Lange WC, Uges DR, van der Werf TS, Kosterink JG, Alffenaar JW. Clarithromycin increases linezolid exposure in multidrug-resistant tuberculosis patients. Eur Respir J. 2013 Dec;42(6):1614-21. doi: 10.1183/09031936.00001913. Epub 2013 Mar 21. PMID 23520311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at the Tuberculosis Centre Beatrixoord (University of Groningen, University Medical Center Groningen, Haren, The Netherlands).
  Dates of recruitment: from december 2011 to november 2012.
Pre-assignment Details: Not applicatble.
Groups:
- 0mg, 250mg and 500mg Claritromycin: Patients receive 300mg linezolid twice a day during entire study.
Period: Linezolid Without Clarithromycin (1 wk)
Arm/Group | 0mg, 250mg and 500mg Claritromycin
Started | 7
Completed | 7
Not Completed | 0
Period: Linezolid + 250mg Claritromycin (wk 2&3)
Arm/Group | 0mg, 250mg and 500mg Claritromycin
Started | 7
Completed | 6
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Linezolid + 500mg Claritromycin (wk 4&5)
Arm/Group | 0mg, 250mg and 500mg Claritromycin
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Clarithromycin: Patients receive 300mg linezolid twice a day during entire study. After one week, 250mg claritromycin once daily is added for a duration of two weeks.
  After another two weeks, 250mg claritromycin is replaced by 500mg claritromycin once daily for another two weeks.
  After this, there is a wash-out period of one week during which no claritromycine is administered.
  Addition of different doses of clarithromycin. : At week 1, 250mg clarithromycin once a day will be added to linezolid therapy during two weeks.
  At week 3, 500mg clarithromycin once a day will be added to linezolid therapy during to weeks.
Arm/Group | Clarithromycin
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  Netherlands | 5

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Time Concentration Curve (AUC0-12h) of Linezolid in Plasma After Addition of 0mg, 250mg, or 500mg Clarithromycin (CLA).
Description: The AUCs of linezolid will be measured at 3 time points after addition of 3 different clarithromycin dosages.
  Samples were obtained before doseing and 1h, 2h, 3h, 4h, 8h, and 12h after administration of linezolid (and claritromycin depending on the period).
Time Frame: At week 1 (baseline), week 3 (250mg clarithromycin), and week 5(500mg clarithromycin).
Measure: Median (Inter-Quartile Range); unit: mg*h/L
Groups:
- 0mg Claritrhomycin: Patients receive 300mg linezolid twice a day during entire study. After one week, 250mg claritromycin once daily is added for a duration of two weeks.
  After another two weeks, 250mg claritromycin is replaced by 500mg claritromycin once daily for another two weeks.
  After this, there is a wash-out period of one week during which no claritromycine is administered.
  Addition of different doses of clarithromycin. : At week 1, 250mg clarithromycin once a day will be added to linezolid therapy during two weeks.
  At week 3, 500mg clarithromycin once a day will be added to linezolid therapy during to weeks.
Arm/Group | 0mg Claritrhomycin | 250mg Clarithromycin | 500mg Clarithromycin
Number analyzed (Participants) | 5 | 5 | 5
mg*h/L | 36.3 [33.2 to 46.3] | 61.0 [34.6 to 63.9] | 67.2 [66.9 to 76.0]

2. Secondary Outcome: Linezolid (LIN) and Clarithromycin (CLA) Pharmacokinetic Parameters, e.g. Tmax, Cmax, Cmin, T1/2, Cl.
Time Frame: At week 1 (baseline), week 3 (250mg clarithromycin), and week 5 (500mg clarithromycin) and week 6 (baseline).
Reporting Status: Not Posted

3. Secondary Outcome: Number of Patients With Adverse Events (AEs)
Description: To assess short-term safety and tolerability when combining linezolid (LIN) with clarithromycin (CLA) by monitoring AEs, i.e. gastro-intestinal effects, hyperlactatemia, haematological abnormalities and neuropathy.
Time Frame: Up to week 6
Population: No serious adverse events
Measure: Number; unit: participants
Groups:
- 0mg Claritromycin; 250mg Clarithromycin; 500mg Clarithromycin: Patients receive 300mg linezolid twice a day during entire study. After one week, 250mg claritromycin once daily is added for a duration of two weeks.
  After another two weeks, 250mg claritromycin is replaced by 500mg claritromycin once daily for another two weeks.
  After this, there is a wash-out period of one week during which no claritromycine is administered.
  Addition of different doses of clarithromycin. : At week 1, 250mg clarithromycin once a day will be added to linezolid therapy during two weeks.
  At week 3, 500mg clarithromycin once a day will be added to linezolid therapy during to weeks.
Arm/Group | 0mg Claritromycin | 250mg Clarithromycin | 500mg Clarithromycin
Number analyzed (Participants) | 5 | 5 | 5
participants | 0 | 0 | 0

4. Secondary Outcome: Pharmacokinetic Parameters, e.g. Tmax, T1/2, Cmax, Cmin, Cl, of Anti-TB Drugs That Are Co-administered as Part of the Continued Standard Care.
Time Frame: At week 1 (baseline), week 3 (250mg clarithromycin) and week 5 (500mg clarithromycin)
Reporting Status: Not Posted

5. Secondary Outcome: Area Under the Time Concentration Curve (AUC0-12h) of Linezolid in Saliva.
Description: The data will be used to clinically validate the analysis linezolid in saliva as surrogate marker for linezolid in plasma.
Time Frame: At week 3 (after co-administration of 250mg clarithromycin)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 0mg Claritromycin | 250mg Clarithromycin | 500mg Clarithromycin
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0mg Claritromycin (N=5) | 250mg Clarithromycin (N=5) | 500mg Clarithromycin (N=5)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No